CLINICAL TRIAL: NCT06537206
Title: Effect of Warm Water Foot Bath on Fever Management in Children: A Randomized Controlled Trial
Brief Title: Foot Bath on Fever Management in Children (EWWFBFMC)
Acronym: EWWFBFMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Sermin Dinc, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-2268639050.99-46589
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries

STUDY DESIGN:
Intervention Model Description: Randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Footbath (Experimental): The experimental group will then receive the first foot bath with water at 38-40°C for approximately 10 minutes. After this, the second set of physiological parameters will be measured at the 40th minute. The child will rest for 10 minutes, followed by measurement and recording of the third set of parameters at the 50th minute.
  A second foot bath at 38-40°C will be applied for another 10 minutes. After this, the fourth set of physiological parameters will be measured, and the FLACC pain score (2nd measurement) will be recorded by the same nurse observer and parent at the 60th minute. The procedure will then be terminated.
  Interventions: Other: Application Footbath
- Control Group (No Intervention): Approximately 10 minutes after the application of the antipyretic, the adaptation of the family and the child to the clinic will be awaited. Children and families who meet the sample selection criteria and verbally and in writing agree to participate in the study will be included.
  A data collection form will be applied to all members of the sample group, and the information will be recorded by the researcher on the form. (20th minute) The parents of the children and the observer nurse will be explained how to use the FLACC pain assessment scale. For inter-observer agreement, the nurse administering the antipyretic and the accompanying parent will simultaneously evaluate using the scale. Throughout the process, the parents of both groups will be with the child.

INTERVENTIONS:
Other: Application Footbath — The foot bath application for the experimental group will be applied with water at 38-40 degrees Celsius for an average of 10 minutes under thermometer control. Immediately afterward, the second physiological parameters will be measured.
  Arms: Application Footbath

SUMMARY:
Reducing the dependency on medication in lowering fever, which is one of the most common symptoms in childhood, and developing safer and more feasible alternative methods are important for child health. This study aims to evaluate the effect of warm water foot baths on vital signs and pain in children, and to scientifically investigate this effect through a randomized controlled trial.

DETAILED DESCRIPTION:
Fever is one of the most common symptoms in childhood, especially in children under the age of five. While it is the most frequent reason for visits to healthcare institutions, it accounts for 25% of pediatric emergency visits. Lack of knowledge about fever in parents triggers fear, and the thought that it can cause seizures, disability, and brain damage induces anxiety and panic in many families. In the presence of anxiety and panic, families may quickly resort to early and incorrect treatment. Administering less medication than necessary for low fevers or high doses for high fevers, repeated use of antipyretics, and inappropriate use of antibiotics lead to ineffective management, resulting in an increase in repeated emergency visits and unnecessary crowding in emergency services. Published guidelines on high fever have emphasized focusing on pain and comfort rather than reducing fever in children. It is reported that foot baths, preferred in pain management, effectively reduce pain and increase comfort. Additionally, guidelines related to fever highlight that warm applications after medication administration can effectively lower persistent fever. Warm water foot bath therapy dilates blood vessels, increases blood circulation, releases heat as sweat, and supports increased oxygenation. Increased circulation improves tissue nutrition and reduces stress. Literature has shown that body temperature decreased in children who received a warm water foot bath. Similarly, studies reported that warm water foot baths were effective in reducing fever in individuals with complaints of high fever.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 1-5 years old. The child has presented to the emergency department with a fever of 38.3°C or higher.
* The child is a patient with "Green Area" (specific condition or disease). The child has no chronic illness. The child has not used any other antipyretic medication in the last 6 hours.
* The child has been administered 15 mg/kg of oral paracetamol as prescribed by the doctor.
* The child and their parent(s) have volunteered to participate in the study. Written consent from the parent(s) is obtained.

Exclusion Criteria:

* Individuals who have not agreed to participate voluntarily in the study.
* Children who have been unable to take paracetamol due to spillage or vomiting.
* Children with compromised skin integrity.
* Individuals who have undergone surgical procedures that would hinder the child's activity.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
FLACC SCORE | 0 minute
  Pain Scale (Max 10 Points, Min. 0 Points) 0 points: No Pain. 10 Points: High Pain
FLACC SCORE | 30 minute
  Pain Scale (Max 10 Points, Min. 0 Points) 0 points: No Pain. 10 Points: High Pain
FLACC SCORE | 50 minute
  Pain Scale (Max 10 Points, Min. 0 Points) 0 points: No Pain. 10 Points: High Pain

SECONDARY OUTCOMES:
Heart Rate | 0 minute
  Heart Rate
Heart Rate | 30 minute
  Heart Rate
Heart Rate | 40 minute
  Heart Rate
Heart Rate | 50 minute
  Heart Rate
Heart Rate | 60 minute
  Heart Rate

OTHER OUTCOMES:
Respiration Rate | 0 minute
  Respiration Rates
Respiration Rate | 30 minute
  Respiration Rates
Respiration Rate | 40 minute
  Respiration Rates
Respiration Rate | 50 minute
  Respiration Rates
Respiration Rate | 60 minute
  Respiration Rates
SpO2 | 0 minute
  Saturation Level
SpO2 | 30 minute
  Saturation Level
SpO2 | 40 minute
  Saturation Level
SpO2 | 50 minute
  Saturation Level
SpO2 | 60 minute
  Saturation Level
Fever | 0 minute
  Body Temparature
Fever | 30 minute
  Body Temparature
Fever | 40 minute
  Body Temparature
Fever | 50 minute
  Body Temparature
Fever | 60 minute
  Body Temparature

CONTACTS AND LOCATIONS:
Overall Officials: semin dinç, Principal Investigator — Atlas University
Locations (2):
- Turkey (Türkiye) (2):
  - Atlas Üniversity, Kağıthane, Istanbul
  - Atlas University, Kâğıthane, Istanbul

IPD SHARING:
Plan to Share IPD: No